CLINICAL TRIAL: NCT03727620
Title: Clinical Effects of Doxycycline in the Treatment of Aggressive Periodontitis: Comparative Clinical Study
Brief Title: Doxycycline in the Treatment of Aggressive Periodontitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mohammed V Souissi University (Other)
Responsible Party: Principal Investigator, BENRACHADI Latifa, Professor, Mohammed V Souissi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOXYAPG18
Record Dates: First submitted 2018-10-10; First posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Aggressive Periodontitis
Keywords: aggressive periodontitis; systemic antibiotics; doxycycline
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Amoxicillin; Metronidazole; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- doxycycline group (Experimental): Drug Longamycine 200 mg the first day , then 100 mg per day for 14 days
  Interventions: Drug: Doxycycline
- amoxicillin plus metronidazole group (Active Comparator): Drug Dispamox 500 mg, 3 times a day for 7 days Flagyl 250 mg, 3 times a day for 7 days
  Interventions: Drug: amoxicillin plus metronidazole

INTERVENTIONS:
Drug: amoxicillin plus metronidazole — patients were administered 250 mg of Flagyl and 500 mg of Dyspamox, three times a day for 7 days
  Other Names: Dispamox and Flagyl
  Arms: amoxicillin plus metronidazole group
Drug: Doxycycline — patients were administered 200 mg of Longamycine the first day and 100 mg per day for 14 days
  Other Names: Longamycine
  Arms: doxycycline group

SUMMARY:
The aim of the study was to compare the clinical effects of systemic use of doxycycline to amoxicillin plus metronidazole as adjunctive treatment in nonsurgical debridement of aggressive periodontitis (AgP). Twenty four patients with aggressive periodontitis were enrolled in this clinical study. They all received oral hygiene instruction and full-mouth nonsurgical debridement using manual instruments. The test group received as adjunctive antibiotic treatment 200 mg of doxycycline the first day followed by 100 mg per day during 14 days. The control group received 500 of amoxicillin and 250 of metronidazole, three times a day for 7 days.

DETAILED DESCRIPTION:
This comparative clinical study was conducted in the department of Periodontology, Center for Dental Consultation and Treatment (CDCT), Rabat, Morocco.

Prior to participation, the purpose of the investigation was fully explained to all participants and written informed consent was obtained from all patients. The study protocol was approved by the biomedical ethical committee of University Mohammed V in Rabat, Morocco, and conducted according to the principles outlined in the Declaration of Helsinki on experimentation involving human subjects.

Patients : Twenty four subjects diagnosed with localized (LAgP) or generalized aggressive periodontitis (GAgP) (8 patients with LAgP and 16 with GAgP) were enrolled in the study. Patients were aged between 16 and 26 years and were from both genders (22 female and 2 male).The diagnosis was based on the classification of the American Academy of Periodontology (AAP).

Clinical variables were pocket depth, plaque index, gingival index

At the end of the debridement sessions, patients were assigned doxycycline or the amoxicillin plus metronidazole regardless the type of AgP. So that, experimental group of patients were administered 200 mg of doxycycline the first day followed by 100 mg per day for 14 days, and the control group were administered 250 mg of metronidazole and 500 mg of amoxicillin, three times a day for 7 days.

Data analysis The data were analyzed using the patient as a unit (subject based analysis). The statistical analysis was performed with a statistical program (SPSS Inc., Chicago, IL, USA). The improvement of periodontal status was evaluated by calculating, for each patient, the difference in Plaque Index (DIP), gingival index (DIG) and probing depth (DPD) ≥ 4mm, between baseline and 3 months post treatment. For each patient, the quantitative variables (PI, GI, and MPD) were expressed as medians and quartiles and were compared before and after treatment using the Wilcoxon test. Improved plaque index (DIP), gingival index (DIG), and probing depth (DPD ≥ 4mm) was compared between the two groups (doxycycline and amoxicillin plus metronidazole) using the Mann-Whitney test. A level P<0,05 was accepted for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* subjects in good general health,
* presence of at least 20 teeth,
* no periodontal treatment performed during the previous 12 months,
* absence of antibiotic intake during six months before the study,
* and no known allergies to antibiotics used in the study

Exclusion Criteria:

* pregnancy,
* lactation,
* and smoking.

Ages: 16 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2014-06-06 (Actual); Study Completion 2014-12-08 (Actual)

PRIMARY OUTCOMES:
Decrease of periodontal pockets ≥ 4mm | 3 months
  • Probing pockets depths were assessed to the nearest millimeter using a standard periodontal probe, when recruiting patient at baseline and the re-evaluation 3 months after nonsurgical mechanical debridement.

SECONDARY OUTCOMES:
Plaque index decrease | 3 months
  Plaque index was assessed by using Loe and silness scores at baseline and the re-evaluation 3 months after nonsurgical mechanical debridement
Gingival index decrease | 3 months
  Gingival index was assessed by using Loe and silness scores at baseline and and at the re-evaluation 3 months after nonsurgical mechanical debridement

CONTACTS AND LOCATIONS:
Overall Officials: Latifa BENRACHADI, Professor, Principal Investigator — Faculty of medicine dentistery, Mohammed V University of Rabat
Locations (1):
- BENRACHADI Latifa, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrera D, Sanz M, Jepsen S, Needleman I, Roldan S. A systematic review on the effect of systemic antimicrobials as an adjunct to scaling and root planing in periodontitis patients. J Clin Periodontol. 2002;29 Suppl 3:136-59; discussion 160-2. doi: 10.1034/j.1600-051x.29.s3.8.x. PMID 12787214
- [Background] Guerrero A, Nibali L, Lambertenghi R, Ready D, Suvan J, Griffiths GS, Wilson M, Tonetti MS. Impact of baseline microbiological status on clinical outcomes in generalized aggressive periodontitis patients treated with or without adjunctive amoxicillin and metronidazole: an exploratory analysis from a randomized controlled clinical trial. J Clin Periodontol. 2014 Nov;41(11):1080-9. doi: 10.1111/jcpe.12299. Epub 2014 Sep 11. PMID 25139116
- [Background] Xajigeorgiou C, Sakellari D, Slini T, Baka A, Konstantinidis A. Clinical and microbiological effects of different antimicrobials on generalized aggressive periodontitis. J Clin Periodontol. 2006 Apr;33(4):254-64. doi: 10.1111/j.1600-051X.2006.00905.x. PMID 16553634